CLINICAL TRIAL: NCT00555412
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Staccato® Loxapine for Inhalation in Subjects on Chronic, Stable Antipsychotic Regimens
Brief Title: Staccato Loxapine Multidose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: Atlanta Center for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-102
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2013-06

CONDITIONS: Volunteers on Chronic, Stable Antipsychotic Regimens
Keywords: pharmacokinetic; multidose; Staccato Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A - 10 mg loxapine q 4 h x 3 (30 mg total) (Experimental)
  Interventions: Drug: A - 10 mg loxapine q 4 h x 3 (30 mg total)
- B - 10 mg x 1, 5 mg x 2 loxapine q 4 h (20 mg total) (Experimental)
  Interventions: Drug: B - 10 mg x 1, 5 mg x 2 loxapine q 4 h (20 mg total)
- C - 5 mg loxapine q 4 h x 3 (15 mg total) (Experimental)
  Interventions: Drug: C - 5 mg loxapine q 4 h x 3 (15 mg total)
- D - inhaled placebo q 4 h x 3 (Placebo Comparator)
  Interventions: Drug: D - inhaled placebo q 4 h x 3

INTERVENTIONS:
Drug: A - 10 mg loxapine q 4 h x 3 (30 mg total) — loxapine aerosol inhalation high dose regimen (30 mg total)
  Other Names: Staccato Loxapine 10 mg
  Arms: A - 10 mg loxapine q 4 h x 3 (30 mg total)
Drug: B - 10 mg x 1, 5 mg x 2 loxapine q 4 h (20 mg total) — loxapine aerosol inhalation middle dose regimen (20 mg total)
  Other Names: Staccato Loxapine 5 and 10 mg
  Arms: B - 10 mg x 1, 5 mg x 2 loxapine q 4 h (20 mg total)
Drug: C - 5 mg loxapine q 4 h x 3 (15 mg total) — loxapine aerosol inhalation low dose regimen (15 mg total)
  Other Names: Staccato Loxapine 5 mg
  Arms: C - 5 mg loxapine q 4 h x 3 (15 mg total)
Drug: D - inhaled placebo q 4 h x 3 — placebo aerosol inhalation (0 mg total)
  Other Names: Staccato Placebo
  Arms: D - inhaled placebo q 4 h x 3

SUMMARY:
The objectives of this trial are to assess the safety, tolerability, and pharmacokinetics of multiple inhaled doses of Staccato Loxapine.

DETAILED DESCRIPTION:
The purpose of the present Phase 1 study in schizophrenic patients is to assess the safety and pharmacokinetics of multiple doses of Staccato Loxapine given within a 24 hour time period. The study will be conducted in schizophrenic patients who are on chronic, stable antipsychotic medication. Patients meeting entry criteria will be randomized to one of three dose sequences of Staccato Loxapine or to Staccato Placebo. Following administration of medications, safety, tolerability and pharmacokinetic assessments will be conducted at serial time points.

ELIGIBILITY:
Inclusion Criteria include:

1. Male and female subjects between the ages of 18 to 65 years, inclusive.
2. Subjects who are on stable, oral, chronic (>2 mos) antipsychotic medication regimen and who are able to tolerate the rapid oral dose taper and substitution regimen.

Exclusion Criteria include:

1. Subjects who are currently treated with injectable depot neuroleptics within one dose interval must be excluded.
2. Subjects who have received loxapine or amoxapine within the last 30 days must be excluded.
3. Subjects with a history of allergy or intolerance to dibenzoxazepines (loxapine and amoxapine) must be excluded.
4. Subjects with a history of movement disorders including Parkinson's disease or a history of neuroleptic malignant syndrome must be excluded.
5. Subjects who have a history within the past year of drug or alcohol dependence or abuse as defined by DSM-4 must be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
PK parameters: tmax, Cmax, AUClast, AUCinf, ke, t1/2 and clearance will be estimated for each subject and for the population using noncompartmental methods. | 48 hours

SECONDARY OUTCOMES:
Plasma concentration-time (PK) profiles will be produced for each subject and a mean PK profile for subjects completing for each dose group | 24 hours
Tolerability will be assessed based on treatment emergent adverse events, vital signs, ECG and a visual-analog sedation scale. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riesenberg, MD, Principal Investigator — Atlanta Center for Medical Research
Locations (1):
- Atlanta Center for Medical Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Spyker DA, Riesenberg RA, Cassella JV. Multiple dose pharmacokinetics of inhaled loxapine in subjects on chronic, stable antipsychotic regimens. J Clin Pharmacol. 2015 Sep;55(9):985-94. doi: 10.1002/jcph.502. Epub 2015 May 6. PMID 25808074